CLINICAL TRIAL: NCT00552409
Title: Randomized Controlled Trial of Vitamin D3 in Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Washington Institute for Translational Health Science (KL2) (Other)
Responsible Party: Principal Investigator, Ian deBoer, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31615-D; 1KL2RR025015-01 (NIH); 5P30DK017047 (NIH); 07-5221-A 01
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus; Chronic Kidney Disease; Diabetic Kidney Disease
Keywords: Diabetes mellitus; Type 2 diabetes; Chronic kidney disease; Diabetic kidney disease; Microalbuminuria; Albuminuria; Vitamin D; Cholecalciferol; Kidney; Renal; Cardiovascular; Clinical trial; Placebo
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Diabetic Nephropathies; Diabetes Mellitus, Type 2; Albuminuria | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Experimental)
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 2000 IU by mouth daily for one year
  Arms: Cholecalciferol
Dietary Supplement: Placebo — One softgel daily for one year
  Arms: Placebo

SUMMARY:
This study will assess the effects of vitamin D3 supplementation (cholecalciferol; 2000 IU daily) on serum calcium levels, circulating vitamin D levels, and markers of kidney disease and cardiovascular risk among people with diabetes mellitus and early kidney disease. Eligibility criteria include type 2 diabetes and stage 1-2 chronic kidney disease, defined by a urine albumin-creatinine ratio 30-300 mg/g and an estimated glomerular filtration rate ≥ 60 mL/min. Participants will be randomly assigned to treatment with vitamin D3 or placebo, each taken by mouth once daily for a study duration of one year. Study medications will be added to standard treatment, including an angiotensin converting enzyme inhibitor and/or angiotensin II receptor blocker. We hypothesize that vitamin D3, compared with placebo: (1) is well-tolerated and safe among people with diabetes and kidney disease; (2) results in adequate attained circulating vitamin D levels; and (3) positively affects markers of kidney disease and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* Urine albumin-creatinine ratio 30-1000 mg/g
* Estimated glomerular filtration rate greater than or equal to 60 mL/min
* Treatment with angiotensin converting enzyme inhibitor and/or angiotensin II receptor blocker for greater than or equal to 6 months, with a stable dose for greater than or equal to 3 months
* Blood pressure less than 140/90 (assessed while taking medications)
* Hemoglobin A1c less than 9% (assessed while taking medications)
* 25-hydroxyvitamin D less than 30 ng/mL

Exclusion Criteria:

* Prior dialysis or kidney transplantation
* Known cause of albuminuria other than diabetes
* Planning to leave the area within 12 months
* Life expectancy less than 12 months
* Participation in another clinical trial within 6 months
* Osteoporosis or other established indication for vitamin D therapy
* Vitamin D3 supplement intake greater than 400 IU/day at screening visit
* History of nephrolithiasis
* Serum calcium greater than 10.2 mg/dL
* Dementia, not fluent in English, or unable to provide informed consent without proxy respondent
* Incontinent of urine
* Failure to take greater than or equal to 80% of placebo pills during study run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian H de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Best CM, Riley DV, Laha TJ, Pflaum H, Zelnick LR, Hsu S, Thummel KE, Foster-Schubert KE, Kuzma JN, Cromer G, Larson I, Hagman DK, Heshelman K, Kratz M, de Boer IH, Hoofnagle AN. Vitamin D in human serum and adipose tissue after supplementation. Am J Clin Nutr. 2021 Jan 4;113(1):83-91. doi: 10.1093/ajcn/nqaa295. PMID 33184642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-three participants from medical clinics associated from the University of Washington (Seattle, WA) provided informed consent for this study between February, 2008 through June, 2009.
Pre-assignment Details: Of the 93 participants who provided informed consent, 63 were ineligible, 8 withdrew prior to randomization, and 22 were randomized to treatment.
Period: Overall Study
Arm/Group | Cholecalciferol | Placebo
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 61 (13) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Albumin Excretion
Description: Albumin and creatinine concentrations were measured in 24hr urine collections at baseline, 3 months after randomization, and one year after randomization. We analyzed the difference in log-transformed albumin-creatinine ratio (ACR, mg/g) after randomization (3 months and one year, analyzed together with all available data included) compared with baseline, by treatment assignment. Results are transformed to present percent difference in urine ACR.
Time Frame: Baseline, 3 months, and one year
Population: All participants were analyzed
Measure: Mean (95% Confidence Interval); unit: percent difference
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 11 | 11
percent difference | -21 [-50 to 23] | -5 [-40 to 49]
Statistical Analysis 1: Comparison: Cholecalciferol vs Placebo; Test type: Superiority or Other; Regression, Linear; Mean Difference (Final Values) = -17, 95% CI 2-sided [-56 to 251] — Mean urine ACR on treatment was 17% lower among participants assigned to cholecalciferol, compared to participants assigned to placebo, adjusted for baseline values

ADVERSE EVENTS:
Arm/Group | Cholecalciferol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/11 | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol (N=11) | Placebo (N=11)
sinus infection (Infections and infestations) | 0 (0) | 1 (1)
carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
frozen shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ovarian cyst (General disorders) | 0 (0) | 1 (1)
vaginitis (Infections and infestations) | 0 (0) | 1 (1)
sleep apnea (General disorders) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
toe amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
dizziness (General disorders) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 0 (0) | 1 (2)
edema (General disorders) | 1 (2) | 1 (1)
elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
low blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
lack of energy (General disorders) | 0 (0) | 1 (1)
decreased mood (Psychiatric disorders) | 1 (1) | 1 (1)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
anhedonia (Psychiatric disorders) | 0 (0) | 1 (1)
burned throat (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
cough (General disorders) | 3 (3) | 0 (0)
ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
rash (General disorders) | 2 (2) | 0 (0)
dyspnea (General disorders) | 0 (0) | 1 (1)
abdominal swelling (General disorders) | 1 (3) | 0 (0)
glaucoma (Eye disorders) | 1 (1) | 0 (0)
multiple sclerosis flair (Immune system disorders) | 1 (2) | 0 (0)
cellulitis (Infections and infestations) | 1 (2) | 0 (0)
endovenous laser treatment (General disorders) | 1 (1) | 0 (0)
trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes